CLINICAL TRIAL: NCT04879862
Title: Inter-System Closed-Loop Control of Locomotor and Bladder Function in Individuals With Acute Spinal Cord Injury
Brief Title: Locomotor and Bladder Function in Individuals With Acute Spinal Cord Injury
Acronym: MC-PP-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Angeli (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Claudia Angeli, Associate Professor, Kessler Foundation
Organization: Kessler Foundation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-1024 MC-PP-3; 1UH3NS116238 (NIH)
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
Keywords: locomotion; epidural stimulation; bladder function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The first 8 participants will be assigned to a group. Once technology is developed the last 8 participants will be randomized to a group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Locomotion (Experimental): Participants will receive 160 locomotor training sessions with epidural stimulation. These sessions may occur once a day (stand and step will alternate days) or twice a day (stand and step on the same day) as recommended by the study physician. Participants will train 5 days per week and each session will last between 1 to 1.5 hours.
  Interventions: Combination Product: Epidural stimulation + Stand Training; Combination Product: Epidural stimulation + Step Training
- Bladder+Locomotion (Experimental): Participants will receive 80 sessions of bladder training alone followed by 80 sessions of locomotor training sessions with epidural stimulation. They will be asked to continue with your bladder training once you start locomotor training. Locomotor Training sessions may occur once a day (stand and step will alternate days) or twice a day (stand and step on the same day) as recommended by the study physician. Participants will train 5 days per week and each session will last between 1 to 1.5 hours.
  Interventions: Combination Product: Epidural stimulation + Stand Training; Combination Product: Epidural stimulation + Step Training; Combination Product: Epidural stimulation + Bladder Capacity Training; Combination Product: Epidural stimulation + Bladder Voiding Efficiency Training

INTERVENTIONS:
Combination Product: Epidural stimulation + Stand Training — Participants may use a standing apparatus or a less assistive device such as walker or cane. In case of upper limbs and trunk control insufficient for safely using the standing apparatus, participants will be placed on the treadmill, and a body weight support system. In this case, the level of body weight support will be continuously reduced as the individuals increase their ability to bear weight. A trainer positioned behind the participant will aid in pelvis and trunk stabilization. Trainer(s) positioned at the lower limb will provide manual facilitation for knee extension during standing. Manual facilitation at the trunk-pelvis and at the legs will be used only when needed.Participants will be encouraged to stand for as long as possible throughout the training session, with the goal to stand for 60 minutes with the least amount of assistance.
Combination Product: Epidural stimulation + Step Training — Participants may be placed on the treadmill in an upright position and suspended in a harness. All trainers are careful to provide manual assistance only when needed. A trainer positioned behind the research participant will aid in pelvis and trunk stabilization, as well as appropriate weight shifting and hip rotation during the step cycle. Trainers positioned at each limb will provide manual assistance to promote knee extension and knee flexion and toe clearance. Research participants will step at various body weight load and speed. Research participants will take a break and rest at any time they feel the need to during the session. If independence is achieved during stepping, some training might be performed overground with appropriate assistive device and manual assistance to maintain participant safety. Participants will be encouraged to step for 60 minutes with the least amount of assistance. Seated or standing resting periods will occur when requested by the individuals
Combination Product: Epidural stimulation + Bladder Capacity Training — We will initially conduct daily training for capacity in a supervised on-site lab setting. Optimal configurations will be used. The storage phase configuration will be used until the time for voiding/catheterization. The training procedure will be repeated for up to 8 hours daily on-site until three consecutive stable days of maintaining a consistent capacity values are achieved and deemed safe. In the home setting, participants will record blood pressure values, voided and residual volumes. Participants will return to the lab the following day for monitoring and testing. If assessments show stable outcomes, participants will be allowed to train at home for 7 consecutive days, prior to returning to the lab for clinical evaluation (urodynamics and questionnaires). On the return visit, if their storage/voiding outcomes remained stable over the 7 days, they will be able to start the home-based training for bladder capacity.
  Arms: Bladder+Locomotion
Combination Product: Epidural stimulation + Bladder Voiding Efficiency Training — We will conduct training for voiding efficiency in a supervised on-site lab setting while the participant continues his/her training for capacity. Voiding without catheterization will be attempted. The training procedure will be repeated for up to 8 hours on-site until three stable days of maintaining a consistent voiding efficiency are achieved and deemed safe. The participant will be sent home for one day to perform the stimulation at home. In the home setting, participants will record blood pressure values, voided and residual volumes. Participants will return to the lab the following day for monitoring and testing. If assessments show stable outcomes, participants will be allowed to train at home for 7 consecutive days, prior to returning to the lab for clinical evaluation and questionnaires. On the return visit, if their storage/voiding outcomes remained stable over the 7 days, they will be able to start the home program integrating bladder training for capacity and voiding
  Arms: Bladder+Locomotion

SUMMARY:
The loss of movement and walking ability significantly affects quality of life after spinal cord injury. In addition, bladder dysfunction consistently ranks as one of the top disorders affecting quality of life after spinal cord injury. The overall objective of this study is to demonstrate that epidural stimulation may be a method for improving stepping, standing and bladder function in individuals with spinal cord injury. With the use of epidural stimulation, the investigators propose to investigate how well the participant can stand and walk and how well the participant's bladder can store or hold urine as well as void or empty urine. The results of this study may aid in the development of treatments to help individuals with spinal cord injuries that are unable to stand or walk and have impaired bladder function.

DETAILED DESCRIPTION:
While the investigators have demonstrated the benefits of scES in chronic SCI with one of the largest series (23 patients to date) the investigators are acutely aware of persistent gaps that need to be filled in order to advance the field of neuromodulation forward. Technological advances to upgrade the stimulator's programming and wireless communication platforms are critically needed in order to integrate multiple training paradigms across multiple systems (i.e. motor and autonomic), as well as take advantage of wireless monitoring technology that could improve the patient experience. The extensive patient self-monitoring, for example regular monitoring of blood pressure during bladder filling cycles, and required manual interaction with the programming device to change parameters for optimal stimulation, remains one of the largest limiting factors in the effective utilization of this technology outside of the laboratory. Without technology components developed specifically for individuals with SCI, treatment effects could be lost due to the burden placed on the individual. Our aim is to develop technology that will interact with currently available systems, to facilitate the implementation and integration of training paradigms for the recovery of locomotion and bladder function in individuals with acute SCI and promote safe long-term use of the technology in the home and community. To this end, this study will provide a flexible communication platform specific for SCI, allow for the evaluation of integrated technology in individuals with high plasticity potential (< 1 year post injury) and allow for the longitudinal evaluation of therapeutic benefits of scES as individuals transition from acute to chronic phase of injury.

Aim 1: To evaluate the use of position based sensors internal to the neurostimulator to modulate stimulation parameters used in the training for motor function recovery following severe SCI.

Aim 2: To identify the scES parameters, using physiological feedback (continuous measures of systolic and diastolic pressure and heart rate), that improve bladder storage and emptying while controlling blood pressure following severe SCI.

Aim 3: To improve device technologies and develop predictive learning algorithms that will allow for the integration of multiple training paradigms used by a single participant.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. non-progressive SCI
3. stable medical condition
4. Inability to stand and step independently
5. unable to voluntarily move all individual joints of the legs
6. no current anti-spasticity medication regimen
7. must not have received botox injections in the prior six months
8. Bladder dysfunction as a result of SCI
9. SCI between T1 and T10
10. no greater than 1 year post injury

Exclusion Criteria:

1. ventilator dependent
2. untreated painful musculoskeletal dysfunction, fracture or pressure sore
3. untreated psychiatric disorder or ongoing drug abuse
4. cardiovascular, respiratory, bladder, or renal disease unrelated to SCI
5. pregnant at the time of enrollment or planning to become pregnant during the time course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Ambulation | 80 sessions, approximately 3 months
  Ability to take independent steps
Bladder storage/voiding | 80 sessions, approximately 3 months
  voiding and/or residual volume (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation - Center for Spinal Stimulation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data included in publications will be made accessible to researchers that wish to externally validate our findings in a spreadsheet format. This data will be sent via secure email in a timely manner upon request. Due to the novelty of this intervention, we may restrict the data sharing to outcomes gathered during spinal cord mapping, assessments and certain information about stimulator configuration, secure information about the implant, nor proprietary hardware/software used during training. We will utilize the SCI Common Data Elements (CDEs) developed through the collaboration of the International Spinal Cord Society, the American Spinal Injury Association and the National Institute for Neurologic Disorders and Stroke (NINDS) CDE Projects as the uniform International SCI Data Sets.
Time Frame: Upon request
Access Criteria: Upon request